CLINICAL TRIAL: NCT03110510
Title: SAMSUNG MEDICAL CENTER
Brief Title: FOLFIRI as Salvage Treatment in Metastatic Biliary Tract Cancer (BTC) Patients Who Were Failed After Gemcitabine Containing Chemotherapy: A Phase II Single Arm Prospective Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: institution problem
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-094
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Intervention Model Description: D1 Irinotecan 180 mg/m2 IV D1-2 5-FU 400mg/m2 bolus and then 2400mg/m2 continuous infusion D1 Leucovorin 200 mg/m2 Every 2 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRI (Experimental): D1 Irinotecan 180 mg/m2 IV D1-2 5-FU 400mg/m2 bolus and then 2400mg/m2 continuous infusion D1 Leucovorin 200 mg/m2 Until disease progression, patient's refusal or unacceptable toxicities
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: Fluorouracil — 5FU 400mg/m2 bolus and then 2400mg/m2, continuous infusion D1-2
  Other Names: Adrucil
Drug: Irinotecan Hydrochloride — Irinotecan 180 mg/m2
Drug: leucovorin calcium — Leucovorin 200 mg/m2

SUMMARY:
FOLFIRI as a salvage treatment in metastatic biliary tract cancer (BTC) patients who failed gemcitabine containing chemotherapy

DETAILED DESCRIPTION:
Biliary tract carcinoma (BTC) is rare in the Europe and the United States, but not uncommon in Asia and Latin America. The tumor arises from the ductular epithelium of the biliary tree within the liver (intrahepatic), the extrahepatic ducts (extrahepatic), or the gallbladder. Intrahepatic cancer is steadily increasing in the Western world. BTCs carry a poor prognosis with 1-year survival rate of 25%. Although surgery remains the only curative treatment for BTC, most patients present with advanced disease and die within a few months of diagnosis. While a combination of gemcitabine and platinum agents seems to be a conclusive treatment option as first-line treatment until now, the role or the optimal regimen for second-line treatment has not been established.

Few articles about second line treatment in advanced BTC were reported. French group recently reported the retrospective analysis of FOLFIRI regimen in advanced BTC patients. However, there is no prospective trial of FOLFIRI regimen to evaluate the efficacy and safety in advanced BTC patients.

So we plan this study to evaluate the efficacy and safety of FOLFIRI regimen as a second line treatment in biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

Provision of a signed written informed consent Age ≥ 20 Histologically or cytologically confirmed carcinoma of biliary tract Progression after treatment with first line gemcitabine-based chemotherapy ECOG performance status of 0~2 Measurable lesion per RECIST 1.1 criteria Expected life expectancy ≥ 3months Adequate marrow, hepatic, renal and cardiac functions Negative pregnancy test within 28 days Available archival tissue or fresh biopsy

Exclusion Criteria:

Poor performance statue Previous treatment history of irinotecan Hypersensitivity to irinotecan Other primary cancer except properly treated non-melanoma skin cancer, cured cervix carcinoma in situ and other cured solid tumor without evidence of recurrence after 5 years of curative treatment.

Severe co-morbid illness and/or active infections Any other clinical trial therapeutics within 14 days Any anti-cancer therapy within 3 weeks prior to initiation of study treatment (radiotherapy, systemic chemotherapy) CTCAE grade 2 or more adverse events remained Intestinal obstruction or CTCAE grade 3-4 upper GI bleeding within 4 weeks QTcB > 480msec or family history of QT prolongation Current heart problem such as: pooly controlled hypertension cardiomyopathy, clinically significant valvular heart disease, uncontrolled angina, acute coronary syndrome within 6 months.

Severe, uncontrolled systemic disease, active infection such as HBV, HCV or HIV, active bleeding tendency or history of organ transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Overall Overall Response Rate | 15 months

SECONDARY OUTCOMES:
Progression-free survival | 24 months
Overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: joonoh park, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea